CLINICAL TRIAL: NCT02837627
Title: Effect of Different Modalities of Enteral Tube Feeding (ETF) on Gastroesophageal Reflux (GER) in Symptomatic Preterm Infants
Brief Title: Effect of Tube Feeding on Gastroesophageal Reflux in Preterm Infants
Acronym: FT-GER-SO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Ospedale dei Bambini "V. Buzzi", Milano (Unknown)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, Responsible of the Neonatal Intensive Care Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2016-TF
Record Dates: First submitted 2016-02-07; First posted 2016-07-19 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Reflux
Keywords: gastroesophageal reflux; tube enteral feeding; preterm infants
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Tube feeding — During the study period, enteral feeds will be administered according to different tube feeding modalities: bolus feeding followed by the removal of the feeding tube; bolus tube feeding with permanence of the feeding tube for the whole post-prandial period; continuous feeding over a 3-hour period.

SUMMARY:
Due to several promoting factors, gastro-esophageal reflux (GER) is very frequent in preterm infants. To limit the potentially harmful widespread of pharmacological treatment, a step-wise approach, which firstly undertakes conservative strategies, is currently considered the best choice to manage GER in the preterm population. Among the most common conservative strategies, postural measures seem to effectively reduce GER features in symptomatic preterm babies, whereas feed thickening is almost ineffective.

Due to their prematurity, preterm infants <34 weeks gestation are often unable to coordinate sucking, swallowing and breathing, thus requiring a feeding tube to ensure adequate enteral intakes. Continuous feeding and boluses are the most common techniques of enteral tube feeding in Neonatal Intensive Care Units; at present, however, the effects of these techniques on GER features have not been clearly established.

This observational, prospective and explorative study primarily aims to evaluate the effect of different techniques of enteral tube feeding on GER frequency and features in symptomatic preterm infants (gestational age ≤33 weeks) undergoing a diagnostic combined pH and multiple intraluminal impedance (pH-MII) for GER evaluation.

DETAILED DESCRIPTION:
Due to several promoting factors related to the physiological immaturity of the gastro-intestinal tract, gastro-esophageal reflux (GER) is a frequent condition among preterm infants.

GER clinical presentation may vary within a wide range of symptoms, being vomiting, regurgitations and cardiorespiratory events the most common in the preterm population.

Combined pH and multiple intraluminal impedance (pH-MII) is currently considered the best choice for GER diagnosis in preterm infants. While pH monitoring is limited to the detection of acid reflux, combined pH-MII effectively identifies both acid and non-acid GER, which is predominant in preterm infants. Moreover, it allows to evaluate the height reached by the refluxate within the esophageal lumen and to distinguish retrograde fluid bolus movements (reflux) from the anterograde ones (swallows).

In the last decade, GER pharmacological treatment has increasingly widespread in Neonatal Intensive Care Units (NICUs). The provision of anti-histamine2 blockers and proton pump inhibitors in the preterm population, however, might lead to such adverse effects as an increased incidence of necrotizing enterocolitis and infections. Hence, to avoid a useless and potentially harmful pharmacological overtreatment, a step-wise approach, firstly promoting conservative strategies, is currently considered the most advisable choice for GER management in symptomatic preterm infants.

Postural and dietary interventions are the most common conservative strategies and their efficacy in improving GER symptoms and features has been largely investigated.

As previously assessed by pH-MII, both prone and left-side positions were more effective than the right-side or supine ones to significantly improve both acid and non-acid GER features.

Feed thickening is widely employed to reduce vomiting and regurgitations in symptomatic term infants; with regard to the preterm population, however, little data is currently available. The efficacy of thickened fortified human milk on preterm infants with GER symptoms has been previously investigated, observing no benefits. Furthermore, standard human milk fortification itself has been shown to increase GER frequency in preterm infants.

With regard to anti-regurgitation (AR) formulas, the effectiveness of a specific AR formula, thickened with amylopectin and specifically tailored for preterm infants' nutritional needs, has been recently evaluated; the tested thickened formula effectively reduced the number of acid GERs, but no difference was observed in the frequency of non-acid GERs and in the mean esophageal acid exposure, which is known to be the main determinant for the development of gastro-esophageal reflux disease (GERD). Thus, according to these data, feed thickening seem to be almost ineffective in improving GER symptoms and features in preterm infants.

Due to their prematurity, preterm infants <34 weeks gestation are unable to coordinate sucking, swallowing and breathing; thus, to ensure adequate enteral intakes, they are usually fed via an intragastric tube. Continuous and bolus feeding are the most common techniques of enteral tube feeding in NICU settings.

The latter is shown to stimulate cyclical surges of gastrointestinal hormones, thus being considered more physiological. It entails the administration of the meal by gravity or through an infusion pump for a total duration of about 10 minutes, after which the feeding tube could be removed. However, the short time elapsing between the tube insertion for bolus administration and its subsequent removal might provoke a vagal response, characterized by bradycardia and temporary reduction of cardiac output. Moreover, the rapid gastric distension following bolus administration could increase the pressure of lower esophageal sphincter (LES), thus contributing to the refluxate of gastric contents into the esophageal lumen.

On the other hand, continuous feeding allows administering enteral feeds over a longer period (e.g. 2 or 3 hours), at a slower flow rate. It has been associated with better absorption of nutrients and faster gastric emptying, thus it may be preferable in case of delayed gastric motility, gastric residuals and abdominal distension. Moreover, its slow rate of infusion prevents a rapid gastric distension; however, this feeding method requires the permanence of the feeding tube through the LES for the whole feeding period, and this could predispose to the occurrence of gastro-esophageal reflux.

The effect of bolus and continuous feeding on cardio-respiratory events, which could represent clinical atypical manifestations of GER, has been recently evaluated, observing a slight but significant increase of apneic episodes during continuous feeding.

A recent systematic review has aimed to evaluate which of these tube-feeding methods could be more suitable in low birth weight infants with GER symptoms; however, current data are scarce and controversial and do not allow to draw any definitive conclusion.

The aim of this study is to evaluate the effect of different enteral tube feeding modalities, such as bolus and continuous feeding, on pH-MII GER features in tube-fed preterm infants ≤33 weeks gestation, undergoing a diagnostic pH-MII evaluation.

Overall, thirty preterm infants ≤33 weeks gestation will be enrolled if suffering from moderate/severe GER symptoms and if a diagnostic 24-hour pH-MII monitoring has been scheduled to evaluate GER features, according to our clinical practice.

During the 24-h pH-MII monitoring, each infant will receive his meals (usually 8) according to the following sequence:

* 1st meal: optional modality (not considered for statistical analysis);
* 2nd meal: continuous feeding over 3 hours;
* 3rd meal: bolus feeding; the feeding tube remains in place for the whole post-prandial period;
* 4th meal: bolus feeding; the feeding tube is removed after feed administration;
* 5th: continuous feeding over 3 hours;
* 6th : bolus feeding; the feeding tube remains in place for the whole post-prandial period;
* 7th: bolus feeding; the feeding tube is removed after feed administration;
* 8th: optional modality (not considered for statistical analysis). Healthcare assistants will inspect the correct application of this sequence.

The pH-MII device in use for this study (Comfortec pH-MII Sandhill Scientific®) is a nasogastric probe with seven rings, composed by six dipolar impedance channels and one antimony electrode responsible for pH detection and placed in the middle of the distal impedance dipole. Due to these characteristics, pH-MII is able to measure the esophageal height reached by refluxate and to identify the direction of esophageal bolus movements, thereby distinguish between a retrograde flow (reflux) and an anti-retrograde flow (swallow).

The distance between the infant's nose and LES will be determined with Strobel's formula: [baby length (cm) x 0.252 + 5)] - 13%. After placement, the probe's position will be radiographically confirmed.

Data from the pH-MII recording will be automatically acquired on a portable Sleuth Sandhill Scientific system and then stored in a personal computer containing a specific software (BioVIEW Analysis Sandhill Scientific, version 5.0.9). Data analysis will be performed by the aforementioned software and confirmed by direct visual evaluation.

Statistical analysis will be performed by SPSS 20 (Statistical Package for the Social Sciences, SPSS Inc., Chicago, IL, USA) for Windows. Differences between the different modalities in terms of GER frequency and features will be tested by Friedman test (level of significance: p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (≤ 33 weeks gestation), able to tolerate at least 100 ml kg-1 day-1 of fortified human milk or standard preterm formula, affected by severe/moderate GER symptoms (recurrent regurgitations, feeding difficulties, failure to thrive and/or post-prandial desaturations), whose usual treatment includes a 24-h pH-MII diagnostic evaluation.
* Need for tube feeding at the time of pH-MII
* Weight ≥ 1100 g at the time of enrollment
* Obtained written parental consent.

Exclusion Criteria:

* Newborns with serious chronic pathology.
* Ongoing pharmacological treatment that could interfere with gastro-enteral motion functions (pro-kinetics) and/or with gastric acidity (H2 antagonists; proton pump inhibitors; sodium alginate).
* Major congenital malformations (e.g. congenital heart diseases, gastrointestinal abnormalities, malformation syndromes).
* Neonatal necrotizing enterocolitis.
* Ongoing infections.
* Patients with severe clinical conditions that can hinder their participation in this trial (e.g. patent ductus arteriosus, intra-ventricular hemorrhage, hemodynamic instability).
* Administration of experimental medication treatments during the previous two weeks.

Ages: 1 Week to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Due to the exploratory nature of this study, at least 30 preterm infants fulfilling the inclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Increase/reduction in the frequency of pH-MII GERs | 24 hours
  changes in the number of acid, non-acid, liquid and gaseous refluxes

SECONDARY OUTCOMES:
Increase/reduction in the duration of pH-MII GERs | 24 hours
  Changes in the duration of GERs recorded
Increase/reduction in the esophageal height reached by MII GERs | 24 hours
  Changes in the height reached by MII GERs

CONTACTS AND LOCATIONS:
Overall Officials: Luigi T Corvaglia, Prof., Principal Investigator — Neonatal Intensive Care Unit, S.Orsola-Malpighi University Hospital, Bologna (Italy)
Locations (2):
- Italy (2):
  - Neonatal Intensive Care Unit of the S.Orsola-Malpighi Hospital, Bologna
  - SC Neonatologia e Terapia Intensiva Neonatale, Ospedale dei Bambini "V. Buzzi", Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dhillon AS, Ewer AK. Diagnosis and management of gastro-oesophageal reflux in preterm infants in neonatal intensive care units. Acta Paediatr. 2004 Jan;93(1):88-93. PMID 14989446
- [Result] van der Pol RJ, Smits MJ, Venmans L, Boluyt N, Benninga MA, Tabbers MM. Diagnostic accuracy of tests in pediatric gastroesophageal reflux disease. J Pediatr. 2013 May;162(5):983-7.e1-4. doi: 10.1016/j.jpeds.2012.10.041. Epub 2012 Dec 7. PMID 23219449
- [Result] Wenzl TG, Moroder C, Trachterna M, Thomson M, Silny J, Heimann G, Skopnik H. Esophageal pH monitoring and impedance measurement: a comparison of two diagnostic tests for gastroesophageal reflux. J Pediatr Gastroenterol Nutr. 2002 May;34(5):519-23. doi: 10.1097/00005176-200205000-00009. PMID 12050578
- [Result] Malcolm WF, Gantz M, Martin RJ, Goldstein RF, Goldberg RN, Cotten CM; National Institute of Child Health and Human Development Neonatal Research Network. Use of medications for gastroesophageal reflux at discharge among extremely low birth weight infants. Pediatrics. 2008 Jan;121(1):22-7. doi: 10.1542/peds.2007-0381. PMID 18166553
- [Result] More K, Athalye-Jape G, Rao S, Patole S. Association of inhibitors of gastric acid secretion and higher incidence of necrotizing enterocolitis in preterm very low-birth-weight infants. Am J Perinatol. 2013 Nov;30(10):849-56. doi: 10.1055/s-0033-1333671. Epub 2013 Jan 28. PMID 23359235
- [Result] Corvaglia L, Ferlini M, Rotatori R, Paoletti V, Alessandroni R, Cocchi G, Faldella G. Starch thickening of human milk is ineffective in reducing the gastroesophageal reflux in preterm infants: a crossover study using intraluminal impedance. J Pediatr. 2006 Feb;148(2):265-8. doi: 10.1016/j.jpeds.2005.09.034. PMID 16492440
- [Result] Corvaglia L, Rotatori R, Ferlini M, Aceti A, Ancora G, Faldella G. The effect of body positioning on gastroesophageal reflux in premature infants: evaluation by combined impedance and pH monitoring. J Pediatr. 2007 Dec;151(6):591-6, 596.e1. doi: 10.1016/j.jpeds.2007.06.014. Epub 2007 Oct 24. PMID 18035136
- [Result] Aceti A, Corvaglia L, Paoletti V, Mariani E, Ancora G, Galletti S, Faldella G. Protein content and fortification of human milk influence gastroesophageal reflux in preterm infants. J Pediatr Gastroenterol Nutr. 2009 Nov;49(5):613-8. doi: 10.1097/MPG.0b013e31819c0ce5. PMID 19633575
- [Result] Corvaglia L, Aceti A, Mariani E, Legnani E, Ferlini M, Raffaeli G, Faldella G. Lack of efficacy of a starch-thickened preterm formula on gastro-oesophageal reflux in preterm infants: a pilot study. J Matern Fetal Neonatal Med. 2012 Dec;25(12):2735-8. doi: 10.3109/14767058.2012.704440. Epub 2012 Jul 13. PMID 22725606